CLINICAL TRIAL: NCT02026895
Title: Virulence of Staphylococcus Lugdunensis in Severe Infections
Acronym: VISLISI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5616
Record Dates: First submitted 2013-12-09; First posted 2014-01-03 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Staphylococcus Lugdunensis; Bacteremia; Endocarditis; Virulence Factors
MeSH Terms: conditions — Bacteremia; Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient with infection by Staphylococcus lugdunensis (Experimental)
  Interventions: Genetic: Genetic blood sample

INTERVENTIONS:
Genetic: Genetic blood sample

SUMMARY:
The main objective is to identify new virulence factors produced by Staphylococcus lugdunensis that can be associated with clinical sign of severe infections and identified symptoms. The methodological approach is based on the comparison between the production of toxins by a given S. lugdunensis isolate classified in patients groups according to the infection clinically defined. Each group will be compared to the presence or not of studied virulence factors. Clinical features associated with toxin activity are not known for S. lugdunensis. This comparative approach is based on the hypotheses that drove to the definition of patient groups and their clinical criteria. However, in the absence of the evident correlation between production of toxins and kind of infection, the statistical evaluation will be completed by a multi-varied analysis. This approach has not been choosen first because of the multiple parameters that undergo during infection that may reveal relationships without true correlation. About the number of included patients in each defined group, if one of them does not reach the expected count, we still might extend inclusions to 3-6 months more. The presence of severe infections without usually defined risk is intriguing. For these last patients, we have planned, after their individual consent to achieve an exome sequencing. The obtained data will be compared to available resources for the human genome. By filtering data through usual protocols, we hope to able to focus onto few genes that evoke specific sensitivity to infections, e.g. severe endocarditis due to S. lugdunensis without defined risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Signed informed consent form
* Proved infection by Staphylococcus lugdunensis: bacteremia, urine tract infection, endocarditis, bone and joint infections, skin and soft tissue infection, deep infection.

Exclusion Criteria:

* Age under 18
* Pregnancy or breastfeeding
* Contamination by Staphylococcus lugdunensis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Presence/absence of virulence factors | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Several groups will be compared considering the presence/absence of virulence factors:
  Bacteriemic VS non bacteriemic, Deep infection VS Skin/mucosal infection, Foreign body infection VS not, Presence of abscess VS not, Sepsis VS no sepsis, Septic embolism VS not, Portal of entry or not
  The following virulence factors will be searched for:
  TSST-1, enterotoxins, leukotoxins, epidermolysins, beta-hemolysins, SCIN-CHIPS, Sbi, Efb, SdrE

SECONDARY OUTCOMES:
Clinical characteristics of infections | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Characteristics of infection: comorbidities (Charlson score) - history of the disease - clinical, cytological , immunological, inflammatory and organ functions parameters - results of additional tests conducted under their care - response to treatment - morbidity and mortality
Whole human transcriptome analysis for selected patients | Genetic blood samples will be analyzed together after the end of inclusion period (18 months)
Genome sequencing of selected strains of Staphylococcus lugdunensis | Genetic blood samples will be analyzed together after the end of inclusion period (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Yves HANSMANN, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, France

REFERENCES:
- [Result] Argemi X, Martin V, Loux V, Dahyot S, Lebeurre J, Guffroy A, Martin M, Velay A, Keller D, Riegel P, Hansmann Y, Paul N, Prevost G. Whole-Genome Sequencing of Seven Strains of Staphylococcus lugdunensis Allows Identification of Mobile Genetic Elements. Genome Biol Evol. 2017 May 1;9(5). doi: 10.1093/gbe/evx077. PMID 28444231
- [Result] Argemi X, Prevost G, Riegel P, Provot C, Badel-Berchoux S, Jehl F, Olivares E, Hansmann Y. Kinetics of biofilm formation by Staphylococcus lugdunensis strains in bone and joint infections. Diagn Microbiol Infect Dis. 2017 Aug;88(4):298-304. doi: 10.1016/j.diagmicrobio.2017.05.002. Epub 2017 May 12. PMID 28529089
- [Result] Argemi X, Matelska D, Ginalski K, Riegel P, Hansmann Y, Bloom J, Pestel-Caron M, Dahyot S, Lebeurre J, Prevost G. Comparative genomic analysis of Staphylococcus lugdunensis shows a closed pan-genome and multiple barriers to horizontal gene transfer. BMC Genomics. 2018 Aug 20;19(1):621. doi: 10.1186/s12864-018-4978-1. PMID 30126366
- [Result] Argemi X, Hansmann Y, Prola K, Prevost G. Coagulase-Negative Staphylococci Pathogenomics. Int J Mol Sci. 2019 Mar 11;20(5):1215. doi: 10.3390/ijms20051215. PMID 30862021